CLINICAL TRIAL: NCT01835028
Title: Multicenter Prospective Study of Low-Flow Low-Gradient Aortic Stenosis (TOPAS Study Phase III)
Brief Title: Multicenter Prospective Study of Low-Flow Low-Gradient Aortic Stenosis (TOPAS Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: University Hospital, Brest (Other)
Responsible Party: Principal Investigator, Philippe Pibarot, Doctor, Laval University
Other Study IDs: MOP-57745
Record Dates: First submitted 2013-04-16; First posted 2013-04-18 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic Stenosis; Low Flow; Low Gradient; Left Ventricle; Echocardiography, Doppler
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample (lithium-heparin, EDTA), Tissue (explanted aortic valves)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Classical Low-Flow, Low-Gradient AS: Observational study in patients with Classical Low-Flow, Low-Gradient Aortic Stenosis and Low LV Ejection Fraction undergoing surgical aortic valve replacement, transcatheter aortic valve replacement, or conservative management:
  I- Baseline visit: Medical history, physical / functional evaluation, blood biomarkers, resting echocardiography, stress echocardiography, aortic valve calcium scoring by computed tomography, myocardial fibrosis by magnetic resonance imaging II- Follow-up: clinical outcomes, physical / functional evaluation, echocardiography, blood biomarkers
  Interventions: Other: Echocardiography; Other: Computed tomography; Other: Magnetic resonance imaging; Other: Blood biomarkers; Other: Stress echocardiography
- Paradoxical Low-Flow, Low-Gradient AS: Observational study in patients with Paradoxical Low-Flow, Low-Gradient Aortic Stenosis and Preserved LV Ejection Fraction undergoing surgical aortic valve replacement, transcatheter aortic valve replacement, or conservative management:
  I- Baseline visit: Medical history, physical / functional evaluation, blood biomarkers, resting echocardiography, stress echocardiography, aortic valve calcium scoring by computed tomography, myocardial fibrosis by magnetic resonance imaging II- Follow-up: clinical outcomes, physical / functional evaluation, echocardiography, blood biomarkers
  Interventions: Other: Echocardiography; Other: Computed tomography; Other: Magnetic resonance imaging; Other: Blood biomarkers; Other: Stress echocardiography

INTERVENTIONS:
Other: Echocardiography — Observational Study using Imaging and Biomarkers
Other: Computed tomography — Observational Study using Imaging and Biomarkers
Other: Magnetic resonance imaging — Observational Study using Imaging and Biomarkers
Other: Blood biomarkers — Observational Study using Imaging and Biomarkers
Other: Stress echocardiography — Observational Study using Imaging and Biomarkers

SUMMARY:
Low-flow, low-gradient (LF-LG) aortic stenosis (AS) may occur with depressed (i.e. Classical LF; CLF) or preserved (i.e. Paradoxical LF; PLF) LV ejection fraction (LVEF) and both situations are amongst the most challenging encountered in patients with valvular heart disease. Although, CLF-LG AS is recognized has an important clinical entity, current ACC/AHA-ESC guidelines however do not provide precise recommendations for clinical management of these patients . PLF-LG AS is a new entity recently described by our group, which is characterized by more pronounced LV concentric remodeling with smaller LV cavity size and a restrictive physiology leading to impaired LV filling, altered myocardial function, and a low-flow state. Up to recently, this entity was often misdiagnosed, leading to underestimation of AS severity and inappropriate delays for aortic valve replacement surgery (SAVR). The two main challenges in patients with CLF- or PLF- LG AS are to distinguish between a true-severe (TS) versus a pseudo-severe (PS) stenosis and to accurately quantify the extent of myocardial impairment. Unfortunately, the traditional resting and stress echocardiographic parameters currently used to assess the severity of valvular and myocardial dysfunction in patients with LF-LG AS are far from being optimal, and as a consequence, quantification of disease severity and therapeutic management may not be appropriate in a substantial proportion of these patients.

THE GENERAL OBJECTIVES of the TOPAS study are to develop and validate new parameters and biomarkers to improve the assessment of stenosis severity and myocardial impairment, the risk-stratification, and the clinical decision making in patients with LF-LG AS and to assess the impact of the different therapeutic strategies on patient outcomes.

DETAILED DESCRIPTION:
Low-flow, low-gradient (LF-LG) aortic stenosis (AS) may occur with depressed (i.e. Classical LF; CLF) or preserved (i.e. Paradoxical LF; PLF) LV ejection fraction (LVEF) and both situations are amongst the most challenging encountered in patients with valvular heart disease. Although, CLF-LG AS is recognized has an important clinical entity, current ACC/AHA-ESC guidelines however do not provide precise recommendations for clinical management of these patients because there is an important lack of data on this condition. PLF-LG AS is a new entity recently described by our group, which is characterized by more pronounced LV concentric remodeling with smaller LV cavity size and a restrictive physiology leading to impaired LV filling, altered myocardial function, and a low-flow state. Up to recently, this entity was often misdiagnosed, leading to underestimation of AS severity and inappropriate delays for aortic valve replacement surgery (SAVR). The two main challenges in patients with CLF- or PLF- LG AS are to distinguish between a true-severe (TS) versus a pseudo-severe (PS) stenosis and to accurately quantify the extent of myocardial impairment. Unfortunately, the traditional resting and stress echocardiographic parameters currently used to assess the severity of valvular and myocardial dysfunction in patients with LF-LG AS are far from being optimal, and as a consequence, quantification of disease severity and therapeutic management may not be appropriate in a substantial proportion of these patients. Furthermore, it remains uncertain which is the optimal timing and mode of treatment (SAVR vs. Transcatheter Aortic Valve Implantation [TAVI] vs. Medical) for the different subsets of patients with LF-LG AS patients (CLF- vs. PLF- LG AS; TS vs. PS AS; absence vs. presence of myocardial contractile reserve etc.) THE GENERAL OBJECTIVES of the TOPAS study are to develop and validate new parameters and biomarkers to improve the assessment of stenosis severity and myocardial impairment, the risk-stratification, and the clinical decision making in patients with LF-LG AS and to assess the impact of the different therapeutic strategies on patient outcomes.

THE SPECIFIC AIMS of the phase III of the TOPAS study are: (1) To obtain and analyze the parameters of stenosis severity and LV functional impairment measured by stress echocardiography (SE), the degree of valvular calcification measured by multidetector computed tomography (CT), the extent of myocardial fibrosis measured by magnetic resonance imaging (MRI), the blood levels of natriuretic peptides and markers of extracellular matrix (ECM) turn-over, and the occurrence of clinical events in a series of 310 patients with CLF-LG AS (210 in TOPAS- I and II + 100 in TOPAS-III) and in a series of 380 patients with PLF-LG AS (80 in TOPAS II + 300 in TOPAS-III). (2) To measure the weight and calcification of the valves explanted from the patients who will undergo SAVR during follow-up in order to corroborate the actual severity of the stenosis. (3) To assess the usefulness of: i) the projected aortic valve area measured by SE to separate TS from PS AS and predict outcomes in PLF-LG AS; ii) the amount of valvular calcium measured by CT to separate TS from PS AS and predict outcomes in CLF- and PLF- LG AS; iii) the myocardial contractile reserve measured by SE, the extent of myocardial fibrosis measured by MRI, and the plasma levels of BNP and ECM biomarkers to predict operative (SAVR) / procedural (TAVI) risk as well as hemodynamic (LV function), functional (DASI and 6-min walk test distance), and clinical (morbidity-mortality) outcomes in CLF- and PLF- LG AS. (4) To compare the different modes of treatment (SAVR, TAVI, Medical), with respect to hemodynamic, functional, and clinical outcomes.

RELEVANCE OF THE STUDY: There have been very few prospective studies performed until now in patients with LF-LG AS and these studies have included a relatively small number of patients, have often used only one imaging modality (Doppler-echo) and a limited number of biomarkers, and they have generally not included the patients with PLF-LG AS. Our prospective study is the first of its kind, as it will use a complementary multimodality imaging approach and it will measure prospectively conventional parameters of disease severity as well as new emerging parameters and biomarkers developed by our team in large prospective series of patients with CLF- and PLF- LG AS. This study shall contribute to improve the diagnostic evaluation and clinical conduct in patients with LF-LG AS. This new knowledge will lead to the establishment of clinical guidelines for the management of these high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* LVEF≤ 40%
* Indexed aortic valve area (AVA) ≤ 0.6 cm²/m²
* Mean transvalvular gradient < 40 mmHg

Exclusion criteria:

* Pregnant or lactating women
* advanced renal failure
* tumor with metastasis

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with moderate to severe aortic stenosis and Low Fow Low Gradiwnt , with Low and preserved Ejection Fraction wil be selected at primary care clinic
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2002-06; Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | Patients will be followed for 5 years, with an average of 3.5 years

SECONDARY OUTCOMES:
30-day mortality (for patients treated by SAVR or TAVR) | Patients will be followed for 5 years, with an average of 3.5 years
cardiovascular mortality | Patients will be followed for 5 years, with an average of 3.5 years
new major cardiovascular events as defined by VARC: myocardial infarction, stroke, vascular complications, and re-hospitalization for heart failure composite end-point of cardiovascular mortality and hospitalization for heart failure | Patients will be followed for 5 years, with an average of 3.5 years
composite end-point of cardiovascular mortality and hospitalization for heart failure | Patients will be followed for 5 years, with an average of 3.5 years

OTHER OUTCOMES:
(1) Stenosis severity: We will use the weight and calcification of the valve explanted at the time of SAVR as a flow-independent marker of stenosis severity | Patients will be followed for 5 years, with an average of 3.5 years
Hemodynamic (LV function) outcome: The outcome variables will be the changes during follow-up in resting and peak stress values of stroke volume, LVEF, longitudinal strain and plasma levels of BNP; LV flow reserve; LV contractile reserve | Patients will be followed for 5 years, with an average of 3.5 years
Functional outcome: Another important objective of treatment is to improve the patient's functional status and quality of life. The outcome variables will be the changes in Duke Activity Score Index and the 6-min walk test distance during follow-up | Patients will be followed for 5 years, with an average of 3.5 years

CONTACTS AND LOCATIONS:
Locations (11):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Viena General Hospital, Vienna, Austria
- CHU Start Tilman, Liège, Belgium
- Canada (3):
  - Ottawa Heart Institute University, Ottawa, Ontario
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec
  - St Paul's Hospital, Vancouver, Vancouver
- France (3):
  - Hôpital La Timone, Marseille
  - Hôpital Bichat, Paris
  - CHU, Rennes, Rennes
- University Hospital, Münster, Germany

REFERENCES:
- [Background] Blais C, Dumesnil JG, Baillot R, Simard S, Doyle D, Pibarot P. Impact of valve prosthesis-patient mismatch on short-term mortality after aortic valve replacement. Circulation. 2003 Aug 26;108(8):983-8. doi: 10.1161/01.CIR.0000085167.67105.32. Epub 2003 Aug 11. PMID 12912812
- [Background] Mohty D, Dumesnil JG, Echahidi N, Mathieu P, Dagenais F, Voisine P, Pibarot P. Impact of prosthesis-patient mismatch on long-term survival after aortic valve replacement: influence of age, obesity, and left ventricular dysfunction. J Am Coll Cardiol. 2009 Jan 6;53(1):39-47. doi: 10.1016/j.jacc.2008.09.022. PMID 19118723
- [Background] Hachicha Z, Dumesnil JG, Bogaty P, Pibarot P. Paradoxical low-flow, low-gradient severe aortic stenosis despite preserved ejection fraction is associated with higher afterload and reduced survival. Circulation. 2007 Jun 5;115(22):2856-64. doi: 10.1161/CIRCULATIONAHA.106.668681. Epub 2007 May 28. PMID 17533183
- [Background] Hachicha Z, Dumesnil JG, Pibarot P. Usefulness of the valvuloarterial impedance to predict adverse outcome in asymptomatic aortic stenosis. J Am Coll Cardiol. 2009 Sep 8;54(11):1003-11. doi: 10.1016/j.jacc.2009.04.079. PMID 19729117
- [Background] Pibarot P, Dumesnil JG. Low-flow, low-gradient aortic stenosis with normal and depressed left ventricular ejection fraction. J Am Coll Cardiol. 2012 Nov 6;60(19):1845-53. doi: 10.1016/j.jacc.2012.06.051. Epub 2012 Oct 10. PMID 23062546
- [Background] Dumesnil JG, Pibarot P, Carabello B. Paradoxical low flow and/or low gradient severe aortic stenosis despite preserved left ventricular ejection fraction: implications for diagnosis and treatment. Eur Heart J. 2010 Feb;31(3):281-9. doi: 10.1093/eurheartj/ehp361. Epub 2009 Sep 8. PMID 19737801
- [Background] Dumesnil JG, Pibarot P. Evaluation of aortic stenosis severity: new challenges, new solutions. J Am Soc Echocardiogr. 2011 Sep;24(9):992-4. doi: 10.1016/j.echo.2011.07.011. No abstract available. PMID 21867870
- [Background] Pibarot P, Dumesnil JG. Assessment of aortic stenosis severity: when the gradient does not fit with the valve area. Heart. 2010 Sep;96(18):1431-3. doi: 10.1136/hrt.2010.195149. No abstract available. PMID 20813724
- [Background] Pibarot P, Dumesnil JG. Paradoxical low-flow, low-gradient aortic stenosis adding new pieces to the puzzle. J Am Coll Cardiol. 2011 Jul 19;58(4):413-5. doi: 10.1016/j.jacc.2011.01.057. No abstract available. PMID 21757119
- [Background] Pibarot P, Dumesnil JG. Improving assessment of aortic stenosis. J Am Coll Cardiol. 2012 Jul 17;60(3):169-80. doi: 10.1016/j.jacc.2011.11.078. PMID 22789881
- [Background] Picano E, Pibarot P, Lancellotti P, Monin JL, Bonow RO. The emerging role of exercise testing and stress echocardiography in valvular heart disease. J Am Coll Cardiol. 2009 Dec 8;54(24):2251-60. doi: 10.1016/j.jacc.2009.07.046. PMID 19958961
- [Background] Rodriguez-Gabella T, Nombela-Franco L, Auffret V, Asmarats L, Islas F, Maes F, Ferreira-Neto AN, Paradis JM, Dumont E, Cote M, Jimenez-Quevedo P, Macaya C, Pibarot P, Rodes-Cabau J. Transcatheter Aortic Valve Implantation in Patients With Paradoxical Low-Flow, Low-Gradient Aortic Stenosis. Am J Cardiol. 2018 Aug 15;122(4):625-632. doi: 10.1016/j.amjcard.2018.04.044. Epub 2018 May 17. PMID 30064863
- [Background] Annabi MS, Clisson M, Clavel MA, Pibarot P. Workup and Management of Patients With Paradoxical Low-Flow, Low-Gradient Aortic Stenosis. Curr Treat Options Cardiovasc Med. 2018 May 2;20(6):49. doi: 10.1007/s11936-018-0642-y. PMID 29721704
- [Background] Ribeiro HB, Lerakis S, Gilard M, Cavalcante JL, Makkar R, Herrmann HC, Windecker S, Enriquez-Sarano M, Cheema AN, Nombela-Franco L, Amat-Santos I, Munoz-Garcia AJ, Garcia Del Blanco B, Zajarias A, Lisko JC, Hayek S, Babaliaros V, Le Ven F, Gleason TG, Chakravarty T, Szeto WY, Clavel MA, de Agustin A, Serra V, Schindler JT, Dahou A, Puri R, Pelletier-Beaumont E, Cote M, Pibarot P, Rodes-Cabau J. Transcatheter Aortic Valve Replacement in Patients With Low-Flow, Low-Gradient Aortic Stenosis: The TOPAS-TAVI Registry. J Am Coll Cardiol. 2018 Mar 27;71(12):1297-1308. doi: 10.1016/j.jacc.2018.01.054. PMID 29566812
- [Background] Annabi MS, Touboul E, Dahou A, Burwash IG, Bergler-Klein J, Enriquez-Sarano M, Orwat S, Baumgartner H, Mascherbauer J, Mundigler G, Cavalcante JL, Larose E, Pibarot P, Clavel MA. Dobutamine Stress Echocardiography for Management of Low-Flow, Low-Gradient Aortic Stenosis. J Am Coll Cardiol. 2018 Feb 6;71(5):475-485. doi: 10.1016/j.jacc.2017.11.052. PMID 29406851
- [Background] Dahou A, Clavel MA, Dumesnil JG, Capoulade R, Ribeiro HB, O'Connor K, Mathieu P, Beaudoin J, Larose E, Rodes-Cabau J, Pibarot P. Impact of AVR on LV Remodeling and Function in Paradoxical Low-Flow, Low-Gradient Aortic Stenosis With Preserved LVEF. JACC Cardiovasc Imaging. 2017 Jan;10(1):88-89. doi: 10.1016/j.jcmg.2016.07.009. Epub 2016 Nov 9. No abstract available. PMID 27838305
- [Background] Dahou A, Toubal O, Clavel MA, Beaudoin J, Magne J, Mathieu P, Philippon F, Dumesnil JG, Puri R, Ribeiro HB, Larose E, Rodes-Cabau J, Pibarot P. Relationship Between QT Interval and Outcome in Low-Flow Low-Gradient Aortic Stenosis With Low Left Ventricular Ejection Fraction. J Am Heart Assoc. 2016 Oct 20;5(10):e003980. doi: 10.1161/JAHA.116.003980. PMID 27792655
- [Background] Dahou A, Clavel MA, Capoulade R, Bartko PE, Magne J, Mundigler G, Bergler-Klein J, Burwash I, Mascherbauer J, Ribeiro HB, O'Connor K, Baumgartner H, Senechal M, Dumesnil JG, Rosenhek R, Mathieu P, Larose E, Rodes-Cabau J, Pibarot P. Right ventricular longitudinal strain for risk stratification in low-flow, low-gradient aortic stenosis with low ejection fraction. Heart. 2016 Apr;102(7):548-54. doi: 10.1136/heartjnl-2015-308309. Epub 2016 Jan 13. PMID 26762240
- [Background] Dayan V, Vignolo G, Magne J, Clavel MA, Mohty D, Pibarot P. Outcome and Impact of Aortic Valve Replacement in Patients With Preserved LVEF and Low-Gradient Aortic Stenosis. J Am Coll Cardiol. 2015 Dec 15;66(23):2594-2603. doi: 10.1016/j.jacc.2015.09.076. PMID 26670058
- [Background] Le Ven F, Thebault C, Dahou A, Ribeiro HB, Capoulade R, Mahjoub H, Urena M, Nombela-Franco L, Allende Carrera R, Clavel MA, Dumont E, Dumesnil J, De Larochelliere R, Rodes-Cabau J, Pibarot P. Evolution and prognostic impact of low flow after transcatheter aortic valve replacement. Heart. 2015 Aug;101(15):1196-203. doi: 10.1136/heartjnl-2014-307067. Epub 2015 May 21. PMID 25999587
- [Background] Dahou A, Magne J, Clavel MA, Capoulade R, Bartko PE, Bergler-Klein J, Senechal M, Mundigler G, Burwash I, Ribeiro HB, O'Connor K, Mathieu P, Baumgartner H, Dumesnil JG, Rosenhek R, Larose E, Rodes-Cabau J, Pibarot P. Tricuspid Regurgitation Is Associated With Increased Risk of Mortality in Patients With Low-Flow Low-Gradient Aortic Stenosis and Reduced Ejection Fraction: Results of the Multicenter TOPAS Study (True or Pseudo-Severe Aortic Stenosis). JACC Cardiovasc Interv. 2015 Apr 20;8(4):588-96. doi: 10.1016/j.jcin.2014.08.019. Epub 2015 Mar 26. PMID 25819185
- [Background] Dahou A, Bartko PE, Capoulade R, Clavel MA, Mundigler G, Grondin SL, Bergler-Klein J, Burwash I, Dumesnil JG, Senechal M, O'Connor K, Baumgartner H, Pibarot P. Usefulness of global left ventricular longitudinal strain for risk stratification in low ejection fraction, low-gradient aortic stenosis: results from the multicenter True or Pseudo-Severe Aortic Stenosis study. Circ Cardiovasc Imaging. 2015 Mar;8(3):e002117. doi: 10.1161/CIRCIMAGING.114.002117. PMID 25681417
- [Background] Clavel MA, Berthelot-Richer M, Le Ven F, Capoulade R, Dahou A, Dumesnil JG, Mathieu P, Pibarot P. Impact of classic and paradoxical low flow on survival after aortic valve replacement for severe aortic stenosis. J Am Coll Cardiol. 2015 Feb 24;65(7):645-53. doi: 10.1016/j.jacc.2014.11.047. PMID 25677424
- [Background] Mohty D, Boulogne C, Magne J, Pibarot P, Echahidi N, Cornu E, Dumesnil J, Laskar M, Virot P, Aboyans V. Prevalence and long-term outcome of aortic prosthesis-patient mismatch in patients with paradoxical low-flow severe aortic stenosis. Circulation. 2014 Sep 9;130(11 Suppl 1):S25-31. doi: 10.1161/CIRCULATIONAHA.113.007819. PMID 25200051
- [Background] Clavel MA, Cote N, Mathieu P, Dumesnil JG, Audet A, Pepin A, Couture C, Fournier D, Trahan S, Page S, Pibarot P. Paradoxical low-flow, low-gradient aortic stenosis despite preserved left ventricular ejection fraction: new insights from weights of operatively excised aortic valves. Eur Heart J. 2014 Oct 7;35(38):2655-62. doi: 10.1093/eurheartj/ehu152. Epub 2014 Apr 21. PMID 24755006
- [Background] Mohty D, Magne J, Deltreuil M, Aboyans V, Echahidi N, Cassat C, Pibarot P, Laskar M, Virot P. Outcome and impact of surgery in paradoxical low-flow, low-gradient severe aortic stenosis and preserved left ventricular ejection fraction: a cardiac catheterization study. Circulation. 2013 Sep 10;128(11 Suppl 1):S235-42. doi: 10.1161/CIRCULATIONAHA.112.000031. PMID 24030412
- [Background] Le Ven F, Freeman M, Webb J, Clavel MA, Wheeler M, Dumont E, Thompson C, De Larochelliere R, Moss R, Doyle D, Ribeiro HB, Urena M, Nombela-Franco L, Rodes-Cabau J, Pibarot P. Impact of low flow on the outcome of high-risk patients undergoing transcatheter aortic valve replacement. J Am Coll Cardiol. 2013 Aug 27;62(9):782-8. doi: 10.1016/j.jacc.2013.05.044. Epub 2013 Jun 12. PMID 23770162
- [Background] Clavel MA, Ennezat PV, Marechaux S, Dumesnil JG, Capoulade R, Hachicha Z, Mathieu P, Bellouin A, Bergeron S, Meimoun P, Arsenault M, Le Tourneau T, Pasquet A, Couture C, Pibarot P. Stress echocardiography to assess stenosis severity and predict outcome in patients with paradoxical low-flow, low-gradient aortic stenosis and preserved LVEF. JACC Cardiovasc Imaging. 2013 Feb;6(2):175-83. doi: 10.1016/j.jcmg.2012.10.015. PMID 23489531
- [Background] Williams TE, O'Day DM, Head WS, Robinson RD. Measurements of antifungal levels in corneal tissue: a simplified bioassay for amphotericin B. Graefes Arch Clin Exp Ophthalmol. 1990;228(6):538-40. doi: 10.1007/BF00918487. PMID 2265769
- [Background] Clavel MA, Burwash IG, Mundigler G, Dumesnil JG, Baumgartner H, Bergler-Klein J, Senechal M, Mathieu P, Couture C, Beanlands R, Pibarot P. Validation of conventional and simplified methods to calculate projected valve area at normal flow rate in patients with low flow, low gradient aortic stenosis: the multicenter TOPAS (True or Pseudo Severe Aortic Stenosis) study. J Am Soc Echocardiogr. 2010 Apr;23(4):380-6. doi: 10.1016/j.echo.2010.02.002. PMID 20362927
- [Result] Blais C, Burwash IG, Mundigler G, Dumesnil JG, Loho N, Rader F, Baumgartner H, Beanlands RS, Chayer B, Kadem L, Garcia D, Durand LG, Pibarot P. Projected valve area at normal flow rate improves the assessment of stenosis severity in patients with low-flow, low-gradient aortic stenosis: the multicenter TOPAS (Truly or Pseudo-Severe Aortic Stenosis) study. Circulation. 2006 Feb 7;113(5):711-21. doi: 10.1161/CIRCULATIONAHA.105.557678. PMID 16461844
- [Result] Clavel MA, Webb JG, Rodes-Cabau J, Masson JB, Dumont E, De Larochelliere R, Doyle D, Bergeron S, Baumgartner H, Burwash IG, Dumesnil JG, Mundigler G, Moss R, Kempny A, Bagur R, Bergler-Klein J, Gurvitch R, Mathieu P, Pibarot P. Comparison between transcatheter and surgical prosthetic valve implantation in patients with severe aortic stenosis and reduced left ventricular ejection fraction. Circulation. 2010 Nov 9;122(19):1928-36. doi: 10.1161/CIRCULATIONAHA.109.929893. Epub 2010 Oct 25. PMID 20975002
- [Result] Clavel MA, Fuchs C, Burwash IG, Mundigler G, Dumesnil JG, Baumgartner H, Bergler-Klein J, Beanlands RS, Mathieu P, Magne J, Pibarot P. Predictors of outcomes in low-flow, low-gradient aortic stenosis: results of the multicenter TOPAS Study. Circulation. 2008 Sep 30;118(14 Suppl):S234-42. doi: 10.1161/CIRCULATIONAHA.107.757427. PMID 18824760
- [Result] Bergler-Klein J, Mundigler G, Pibarot P, Burwash IG, Dumesnil JG, Blais C, Fuchs C, Mohty D, Beanlands RS, Hachicha Z, Walter-Publig N, Rader F, Baumgartner H. B-type natriuretic peptide in low-flow, low-gradient aortic stenosis: relationship to hemodynamics and clinical outcome: results from the Multicenter Truly or Pseudo-Severe Aortic Stenosis (TOPAS) study. Circulation. 2007 Jun 5;115(22):2848-55. doi: 10.1161/CIRCULATIONAHA.106.654210. Epub 2007 May 21. PMID 17515464
- [Result] Burwash IG, Lortie M, Pibarot P, de Kemp RA, Graf S, Mundigler G, Khorsand A, Blais C, Baumgartner H, Dumesnil JG, Hachicha Z, DaSilva J, Beanlands RS. Myocardial blood flow in patients with low-flow, low-gradient aortic stenosis: differences between true and pseudo-severe aortic stenosis. Results from the multicentre TOPAS (Truly or Pseudo-Severe Aortic Stenosis) study. Heart. 2008 Dec;94(12):1627-33. doi: 10.1136/hrt.2007.135475. Epub 2008 Apr 1. PMID 18381378
- [Result] Clavel MA, Webb JG, Pibarot P, Altwegg L, Dumont E, Thompson C, De Larochelliere R, Doyle D, Masson JB, Bergeron S, Bertrand OF, Rodes-Cabau J. Comparison of the hemodynamic performance of percutaneous and surgical bioprostheses for the treatment of severe aortic stenosis. J Am Coll Cardiol. 2009 May 19;53(20):1883-91. doi: 10.1016/j.jacc.2009.01.060. PMID 19442889
- [Result] Clavel MA, Rodes-Cabau J, Dumont E, Bagur R, Bergeron S, De Larochelliere R, Doyle D, Larose E, Dumesnil JG, Pibarot P. Validation and characterization of transcatheter aortic valve effective orifice area measured by Doppler echocardiography. JACC Cardiovasc Imaging. 2011 Oct;4(10):1053-62. doi: 10.1016/j.jcmg.2011.06.021. PMID 21999863
- [Result] Clavel MA, Dumesnil JG, Capoulade R, Mathieu P, Senechal M, Pibarot P. Outcome of patients with aortic stenosis, small valve area, and low-flow, low-gradient despite preserved left ventricular ejection fraction. J Am Coll Cardiol. 2012 Oct 2;60(14):1259-67. doi: 10.1016/j.jacc.2011.12.054. Epub 2012 May 30. PMID 22657269
- [Derived] Galli E, Le Ven F, Coisne A, Sportouch C, Le Tourneau T, Lavie-Badie Y, Bernard A, Eicher JC, Dreyfus J, Ternacle J, Baleynaud S, Auffret V, Le Pabic E, Pibarot P, Oger E, Donal E. Randomised study for the Optimal Treatment of symptomatic patients with low-gradient severe Aortic valve Stenosis and preserved left ventricular ejection fraction (ROTAS trial). Heart. 2024 Sep 25;110(20):1223-1230. doi: 10.1136/heartjnl-2024-324224. PMID 39209438
- [Derived] Annabi MS, Cote N, Dahou A, Bartko PE, Bergler-Klein J, Burwash IG, Orwat S, Baumgartner H, Mascherbauer J, Mundigler G, Fukui M, Cavalcante J, Ribeiro HB, Rodes-Cabau J, Clavel MA, Pibarot P. Comparison of Early Surgical or Transcatheter Aortic Valve Replacement Versus Conservative Management in Low-Flow, Low-Gradient Aortic Stenosis Using Inverse Probability of Treatment Weighting: Results From the TOPAS Prospective Observational Cohort Study. J Am Heart Assoc. 2020 Dec 15;9(24):e017870. doi: 10.1161/JAHA.120.017870. Epub 2020 Dec 8. PMID 33289422
- [Derived] Dahou A, Clavel MA, Capoulade R, O'Connor K, Ribeiro HB, Cote N, Le Ven F, Rodes-Cabau J, Dumesnil JG, Mathieu P, Pibarot P. B-Type Natriuretic Peptide and High-Sensitivity Cardiac Troponin for Risk Stratification in Low-Flow, Low-Gradient Aortic Stenosis: A Substudy of the TOPAS Study. JACC Cardiovasc Imaging. 2018 Jul;11(7):939-947. doi: 10.1016/j.jcmg.2017.06.018. Epub 2017 Oct 5. PMID 28917673